CLINICAL TRIAL: NCT06758414
Title: Exploring the Efficacy of Cognitive Behavioral Therapy for Chronic Pain in Veterans With Serious Mental Illness
Brief Title: CBT-CP for Veterans With SMI
Acronym: CP-SMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D5049-R; 1 I01 RX005049-01A2 (Other Grant/Funding Number: VA RRDT)
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Pain; Schizophrenia; Psychotic Disorders; Bipolar Disorder; Affective Disorders, Psychotic
Keywords: Veterans; chronic pain; psychotic disorders; affective disorders, psychotic; cognitive behavioral therapy; ecological momentary assessment
MeSH Terms: conditions — Chronic Pain; Schizophrenia; Psychotic Disorders; Bipolar Disorder; Affective Disorders, Psychotic | interventions — Cognitive Behavioral Therapy; Health

STUDY DESIGN:
Intervention Model Description: The investigators plan to randomize N = 190 Veterans equally into one of two conditions, stratified by serious mental illness (SMI) diagnosis (schizophrenia/schizoaffective disorder; bipolar disorder; major depressive disorder with psychotic feature). The investigators will randomize individuals within stratification groups in permuted blocks, ensuring that the intervention and control samples will be the same size once every block has been randomized. This procedure maximizes statistical power. After completing baseline assessments, participants will be randomized into one of two treatment conditions - Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) or Health & Wellness (H&W), an active control matched for time and attention with CBT-CP. Each intervention consists of 11 weekly, individual sessions that last 45-50 minutes. Participants will remain in their assigned intervention for the duration of the study and will not receive the other intervention.
Who Masked: Outcomes Assessor
Masking Description: Trained RAs blind to condition will administer post-treatment and 6-month follow-up assessments. To preserve the blind, participants will be instructed not to reveal their study condition once randomized. If they do, the RA will make a note indicating when the blind was compromised, and a different RA will complete the assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) (Experimental): Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) will be conducted in accordance with the Cognitive Behavioral Therapy for Chronic Pain: Therapist Manual and the VA Evidence-Based Practice (EBP) roll-out training. CBT-CP consists of a 12-session protocol, including an initial assessment session (BL assessment; Session 1), 10 content-specific sessions (pain education, goal-setting, cognitive and behavioral skill building; Sessions 2-11), and a booster session scheduled approximately one month after the final CBT-CP session (Session 12). Participants randomized to the CBT-CP condition (n = 30) will complete one 60-minute individual session per week. Each CBT-CP session will be led by a trained study interventionist using a manualized curriculum, following a basic structure including review of previous session material, introduction of new information or skills, and discussion of how to implement learned material into a home action plan.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Chronic Pain (CBT-CP)
- Health & Wellness (H&W) (Active Comparator): Health & Wellness (H&W) was developed by VISN 5 MIRECC investigators and consists of psychoeducation on topics related to physical and emotional wellbeing. Its structure is similar to CBT-CP (10 weekly individual 60-minute sessions, no booster session). Each Health & Wellness session will be led by a trained interventionist using a manualized curriculum that includes review of previous session material, introduction of new information, and discussion of a range of health-related topics (physical activity/exercise, nutrition/healthy eating, managing medications and side effects, and addictive behaviors (e.g., substance use, gambling, eating) that do not include pain. Typical sessions include discussion of the impact of the topic on overall health and well-being, identifying benefits and challenges to improving or maintaining health in that area, and strategies to address challenges in that area.
  Interventions: Behavioral: Health & Wellness (H&W)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) — Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) will be conducted in accordance with the Cognitive Behavioral Therapy for Chronic Pain: Therapist Manual and the VA Evidence-Based Practice (EBP) roll-out training. CBT-CP consists of a 12-session protocol, including an initial assessment session (BL assessment; Session 1), 10 content-specific sessions (pain education, goal-setting, cognitive and behavioral skill building; Sessions 2-11), and a booster session scheduled approximately one month after the final CBT-CP session (Session 12). Participants randomized to the CBT-CP condition (n = 30) will complete one 60-minute individual session per week. Each CBT-CP session will be led by a trained study interventionist using a manualized curriculum, following a basic structure including review of previous session material, introduction of new information or skills, and discussion of how to implement learned material into a home action plan.
  Arms: Cognitive Behavioral Therapy for Chronic Pain (CBT-CP)
Behavioral: Health & Wellness (H&W) — Health & Wellness (H&W) was developed by VISN 5 MIRECC investigators and consists of psychoeducation on topics related to physical and emotional wellbeing. Its structure is similar to CBT-CP (10 weekly individual 60-minute sessions, no booster session). Each Health & Wellness session will be led by a trained interventionist using a manualized curriculum that includes review of previous session material, introduction of new information, and discussion of a range of health-related topics (physical activity/exercise, nutrition/healthy eating, managing medications and side effects, and addictive behaviors (e.g., substance use, gambling, eating) that do not include pain. Typical sessions include discussion of the impact of the topic on overall health and well-being, identifying benefits and challenges to improving or maintaining health in that area, and strategies to address challenges in that area.
  Arms: Health & Wellness (H&W)

SUMMARY:
Chronic musculoskeletal pain has a highly negative impact on Veterans, especially those with serious mental illness (SMI). Chronic musculoskeletal pain leads to poorer mental and physical health-related functioning, representing a critical obstacle to rehabilitation and recovery for SMI Veterans. Despite known high prevalence rates of chronic pain in SMI populations, there is little research to evaluate nonpharmacological pain management strategies in this population. This study aims to address this research and clinical gap by testing the efficacy of Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) - a VA evidence-based psychotherapy for chronic pain - in Veterans with SMI and chronic low back pain. The study will primarily evaluate the impact of CBT-CP on pain-related functioning, quality of life, and pain severity. This study will also examine relationships between pain and mental health symptoms, and how these relationships may change with CBT-CP completion.

DETAILED DESCRIPTION:
Project Background: Chronic musculoskeletal pain is one of the most common physical health diagnoses among individuals with SMI. Individuals with SMI and chronic musculoskeletal pain report worse mental and physical health functioning relative to people with other mental or physical health conditions. Despite knowing about high rates of chronic musculoskeletal pain among individuals with SMI; little research has been conducted to further understand the complex relation between pain and psychiatric symptoms and consider the usefulness or appropriateness of current treatment approaches. What is known is problematic: Veterans with SMI are largely not provided options for nonpharmacological pain management strategies, including CBT-CP, and are more likely to be prescribed pain medications that pose unique risks to this population.

Project Objectives: The proposed Merit research will address research and clinical gaps by testing the efficacy of CBT-CP in Veterans with SMI and chronic musculoskeletal pain, notably chronic low back pain. The investigators will complete a large, randomized controlled trial with 190 Veterans, comparing CBT-CP to an active control condition ("Health & Wellness"). The investigators will examine effects of treatment on functioning and pain interference, quality of life, and pain severity. The investigators will evaluate these variables at baseline, post-treatment, and six months post-treatment through both standardized assessment procedures and timepoints; as well as a one-week ecological momentary assessment (EMA) period prior to each assessment timepoint. The EMA data will allow us to examine inter- and intra-variability in pain and related functioning, including its relationship to SMI symptoms, and to evaluate how engagement in CBT-CP may affect pain variability and its relationship to mental health.

Project Methods: This project will include completing a randomized control trial (RCT) with 190 Veteran participants, evaluating impact of CBT-CP versus Health & Wellness on pain-related functioning and interference, quality of life, and pain severity. The investigators will also explore process variables, including physical activity and pain catastrophizing, as well as moderators, including SMI diagnosis and symptom severity along with pain severity at baseline, to see how these variables affect treatment engagement and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic back pain, per medical record
* Have a PEG-3 rating of 4 or greater for pain severity or interference
* Meet criteria for an SMI diagnosis (schizophrenia, schizoaffective disorder, bipolar disorder, major depression with psychosis) per medical record
* 18 years of age or older
* Enrolled in outpatient programming within a VISN 5 health care facility at time of consent
* Have regular access to a telephone
* Capacity to sign informed consent

Exclusion Criteria:

* Are engaging in moderate-to-severe substance use that would impact their ability to participate and/or would require a higher level of care (as determined by treating provider)
* Engagement in individual Cognitive Behavioral Therapy for Chronic Pain (CBT-CP), whether currently or in the past 12 months
* Have a current acute pain condition, medical condition, or limited mobility (i.e., unable to walk one city block) that would interfere with their ability to engage in CBT-CP interventions (e.g., activity pacing/walking program)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2026-02-01 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory-Interference (BPI-INT) | post-treatment (~4 months after randomization); 6-month follow-up (~10 months after randomization)
  The Brief pain Inventory - Interference subscale (BPI-INT) is a 9-item questionnaire measuring pain-relate interference. Respondents answer the degree to which pain interferes with mood/affect and physical activity on a scale from 0 (not at all) to 10 (all the time/completely). An average score is calculated, with a score of >= 4 indicating moderate to severe pain interference. The instrument has excellent psychometric properties and is regularly used in pain research and clinical practice.
Veterans RAND 36-Item Health Survey (VR-36) | post-treatment (~4 months after randomization); 6-month follow-up (~10 months after randomization)
  The Veterans RAND 36-Item Health Survey (VR-36) is a 36-item questionnaire measuring health-related quality of life and 8 domains of health-related functioning (physical functioning, role limitations due to physical problems, role limitations due to emotional problems, bodily pain, general health perceptions, vitality, social functioning, and mental health). Items are scored on a 3- to 6-point scale and are summed to create a total and domain scores, ranging from 0 (worst health status) to 100 (best health status). The VR-36 demonstrated improved reliability, precision, and validity compared to the SF-36 and among persons with SMI.
PEG-3 | post-treatment (~4 months after randomization); 6-month follow-up (~10 months after randomization)
  The PEG-3 will assess pain severity and related functioning and quality of life (enjoyment, general activity), using a 0 to 10 rating scale with qualifying statements for each numeric rating; a rating of 4 or greater indicates moderate-to-severe pain intensity. The PEG-3 will be included in the Ecological Momentary Assessment (EMA) surveys; Veterans will be asked about the extent to which they have experienced each item in the one hour prior to survey completion. The PEG-3 has been validated in Veterans receiving VA primary care services and has good reliability and validity when compared to longer pain assessments. As a primary outcome, changes in the two items assessing functioning (General activity interference) and quality of life (Enjoyment of life) will be examined.

SECONDARY OUTCOMES:
Pain Numeric Rating Scale (PNRS) | post-treatment (~4 months after randomization); 6-month follow-up (~10 months after randomization)
  Pain severity will be rated using the Pain Numeric Rating Scale (PNRS). It is a 3-item scale assessing the person's average, worst, and least pain during the past week. Each item is rated on a scale from 0 (no pain) to 10 (worst pain). The items are averaged together to create a more accurate "average" pain score, with a score of >= 4 indicating moderate to severe pain severity.
PEG-3 | post-treatment (~4 months after randomization); 6-month follow-up (~10 months after randomization)
  The PEG-3 will assess pain severity and related functioning and quality of life (enjoyment, general activity), using a 0 to 10 rating scale with qualifying statements for each numeric rating; a rating of 4 or greater indicates moderate-to-severe pain intensity. The PEG-3 will be included in the Ecological Momentary Assessment (EMA) surveys; Veterans will be asked about the extent to which they have experienced each item in the one hour prior to survey completion. The PEG-3 has been validated in Veterans receiving VA primary care services and has good reliability and validity when compared to longer pain assessments. As a secondary outcome, changes in the Pain severity item will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Letitia Travaglini, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Travaglini LE, Bennett M, Kacmarek CN, Kuykendall L, Coakley G, Lucksted A. Barriers to accessing pain management services among veterans with bipolar disorder. Health Serv Res. 2023 Dec;58(6):1224-1232. doi: 10.1111/1475-6773.14221. Epub 2023 Sep 4. PMID 37667502
- [Background] Travaglini LE, Kuykendall L, Bennett ME, Abel EA, Lucksted A. Relationships between chronic pain and mood symptoms among veterans with bipolar disorder. J Affect Disord. 2020 Dec 1;277:765-771. doi: 10.1016/j.jad.2020.08.069. Epub 2020 Sep 1. PMID 33065815